CLINICAL TRIAL: NCT02633514
Title: A Randomized Phase III Study of Adjuvant Radiotherapy Versus Adjuvant Radiochemotherapy in Patients With Incomplete ResectionThymoma or Thymic Carcinoma
Brief Title: Adjuvant Treatment for Incomplete Resection Thymoma or Thymic Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kailiang Wu, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1508151-6
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Thymoma and Thymic Carcinoma
Keywords: thymoma; thymic carcinoma; adjuvant radiotherapy; adjuvant radiochemotherapy; incomplete resection
MeSH Terms: conditions — Thymoma | interventions — Cisplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiochemotherapy (Experimental): adjuvant radiochemotherapy after incomplete resection: Cisplatin + Etoposide + Radiotherapy (60Gy / 30FX)
  Interventions: Drug: Cisplatin; Drug: Etoposide; Radiation: radiotherapy
- radiotherapy (Sham Comparator): adjuvant radiotherapy after incomplete resection: Radiotherapy (60Gy / 30FX)
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Drug: Cisplatin — 25mg/m2,iv gtt,d1-3
  Other Names: DDP
  Arms: Radiochemotherapy
Drug: Etoposide — 75mg/m2,iv gtt,d1-3
  Other Names: VP-16
  Arms: Radiochemotherapy
Radiation: radiotherapy — 60Gy/30Fx

SUMMARY:
This study is designed to investigate whether adjuvant radiochemotherapy after incomplete resection has a better survival than adjuvant radiotherapy for thymoma or thymic carcinoma.

DETAILED DESCRIPTION:
The previous trials have showed that radiotherapy was significantly associated with prolonged OS and chemotherapy is playing an increasing role in treatment of patients with thymoma or thymic carcinoma.However,whether patients with thymoma or thymic carcinoma could benefit from adjuvant radiochemotherapy after incomplete resection remains controversial. The purpose of this study is to investigate whether adjuvant radiochemotherapy after incomplete resection can improve survival for thymoma or thymic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

18~75 years old; Eastern Cooperative Oncology Group performance status of 0 to 2; Pathologically confirmed ; incomplete resection (R1 or R2);have adequate bone marrow, hepatic, and renal function;Patients receive incomplete resection within 3 months; Written informed consent.

Exclusion Criteria:

Patients with distant metastases; Patients underwent radiotherapy or chemotherapy; Patients who have malignancy history excluding carcinoma in situ of cervix in the previous five years; Active clinical pulmonary infection; Pregnant or nursing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  from registration to disease progression or death.

SECONDARY OUTCOMES:
Overall survival | 2 years
  from registration to death as a result of any cause
Number of Participants with Treatment- Related Adverse Events as Assessed by CTCAE v4.0 | 2 years
  Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Kailiang Wu, MD. PhD, Principal Investigator — Fudan University
Locations (1):
- Kailiang Wu, Shanghai, Shanghai Municipality, China